CLINICAL TRIAL: NCT06552663
Title: The Diagnostic Power Of Coronary Ct Angiography In Patients With Chest Pain And Zero Calcium Score
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Abdellah Farrag Abdelrheim, Resident Doctor, Assiut University
Other Study IDs: Coronary CT Angiography
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: CT - Coronary Thrombosis
MeSH Terms: conditions — Coronary Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CCTA — Coronary CT angiography

SUMMARY:
To prove the non-used wide diagnostic range of CCTA in diagnosis of other causes of chest pain in addition to the traditional known role in coronary atherosclerosis.

DETAILED DESCRIPTION:
The heart is a specialized muscular organ which receives blood via major veins) SVC, IVC ,CS( then pumps it through the arteries (Aorta and Pulmonary artery) towards the systemic and pulmonary circulations. Non oxygenated blood enters the heart via SVC, IVC and CS, passes to the lungs to be oxygenated via the Pulmonary artery then returns to the heart via the Pulmonary veins and finally to the systemic circulation through Aorta.

Cardiac muscles are unique and differs from skeletal and smooth muscles to suit their function, and they are not liable to regenerate like all cells in the body, the cardiac muscles needs to be supplied with oxygen, nutrients and their metabolic wastes must be drained away. This is achieved by the coronary circulation which formed of two main arteries that arise just above the aortic valve, These are the right and left main coronary arteries and their branches. the venous drainage is through the major cardiac veins towards CS that finally drains at the right atrium. [1] As a result any affection of coronary arteries or interruption of blood flow inside it will cause weakness or death of cardiac cells (myocardium).The diseases affecting coronary arteries may be congenital e.g. abnormal course of the coronary arteries or myocardial bridge , traumatic e.g. dissection, inflammatory e.g. Takayasu's arteritis (TAK) , vascular e.g. aneurysm, lastly and the most common is atherosclerosis. [2] Atherosclerosis causes variable degrees of occlusion of the coronary arteries and results in a demand-supply mismatch of oxygen. it typically involves the formation of plaques in the arterial lumen of that impedes blood flow, atherosclerosis may be diffuse (mild subintimal affection), focal or multifocal called atherosclerotic plaques. Plaque is a build-up of fatty material that narrows the vessel lumen and impedes the blood flow, (fatty streak) Which is formed by subendothelial deposition of lipid-laden macrophages (foam cells), smooth muscles and collagen. Over time, this plaque could grow in size or become stable if no further insult occurs to the endothelium. If it becomes stable, a fibrous cap will form, and the lesion will become calcified over time. The drawback of calcified plaque is stenosis that impedes the blood supply while that of soft plaque is liability to further growth, detachment causing arterial occlusion or external rupture causing hemopericardium. [3] So that it is an advantage of CT over coronary catheterization extra coronary lesions either vascular e.g. aortic dissection, pulmonary embolism, cardiac e.g. pericarditis, extracardiac and mediastinal e.g. GERD, or even pleurisy, myositis and other chest pathologies via large FOV scanning through another phase. Cardiovascular diseases do not frequently have symptoms but may cause chest pain which is the most important symptom in CVDs, and may be a sign of other diseases like vascular, inflammatory …etc.

In the past CADs diagnosis could be done by many tests like ECG, blood tests, Cardiac catheterization and angiogram Which is invasive despite of high real time value and ability to place a stent or balloon dilatation. [4] Recently multidetector computed tomography (CT) and CT angiography could be done due to recent equipment that could match the cardiac motion and avoid the artifacts .

A CT scan of the heart can show calcium deposits and blockages in the coronary arteries and be calculated by calcium score, The calcium score is calculated based on the amount of calcification in the vessel walls of coronary arteries observed in a cardiac (CT) scan, Many methods have been used in calcium scoring e.g. Agatston calcium score which is the most popular one. A higher score indicates a larger amount of calcium deposition. However; Ca score of zero is not a sign of negative CVDs, so that CCTA become a must and don't just depend on the coronary Ca score alone.

A CT coronary angiogram is mainly used to check for narrowed or blocked coronary artery by any plaque even the soft non calcified ones . However, it can check for other heart conditions such congenital heart disease, valvular heart disease, carditis, aortic aneurysms…etc.

A CT coronary angiogram differs from a standard coronary angiogram. Which is an invasive technique that could only see the lumen of the artery not the wall itself and calcium score is not available, yet still a real time technique and have a therapeutic value at the same time. [5]

ELIGIBILITY:
Inclusion Criteria:

* patients with chest pain whom are referred by cardiologist for coronary CT angiography and coronary artery calcium score to detect atherosclerosis .

Exclusion Criteria:

* Patients who refuse to sign the consent
* Subjects suspected of having myocardial infarction, unstable angina pectoris, or coronary artery disease
* Subjects who experienced heart attack within 40 days prior to the CT scan
* Subjects with a diagnosed complicated heart anomaly
* BMI > 35 kg/m2
* Serum creatinine ≥ 1.5 mg/dl
* Pregnant subjects
* Subjects with a history of hypersensitivity reaction to contrast agents
* Subjects with contraindications to the use of nitroglycerine
* Subjects who plan to participate or enroll in other randomized clinical trials for cardiovascular disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * community sample
  * primary care clinic
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate outcome of coronary CT angiography in cases with chest pain with zero calcium score . Evaluate outcome of coronary CT angiography in cases with chest pain with zero calcium score . Evaluate outcome of coronary CT angiography | two years
  Evaluate outcome of coronary CT angiography in cases with chest pain with zero calcium score

REFERENCES:
- [Background] Buckberg GD, Nanda NC, Nguyen C, Kocica MJ. What Is the Heart? Anatomy, Function, Pathophysiology, and Misconceptions. J Cardiovasc Dev Dis. 2018 Jun 4;5(2):33. doi: 10.3390/jcdd5020033. PMID 29867011
- [Background] Villa AD, Sammut E, Nair A, Rajani R, Bonamini R, Chiribiri A. Coronary artery anomalies overview: The normal and the abnormal. World J Radiol. 2016 Jun 28;8(6):537-55. doi: 10.4329/wjr.v8.i6.537. PMID 27358682
- [Background] Lusis AJ. Atherosclerosis. Nature. 2000 Sep 14;407(6801):233-41. doi: 10.1038/35025203. PMID 11001066
- [Background] Nelson AJ, Ardissino M, Psaltis PJ. Current approach to the diagnosis of atherosclerotic coronary artery disease: more questions than answers. Ther Adv Chronic Dis. 2019 Nov 1;10:2040622319884819. doi: 10.1177/2040622319884819. eCollection 2019. PMID 31700595
- [Background] Doris M, Newby DE. Coronary CT Angiography as a Diagnostic and Prognostic Tool: Perspectives from the SCOT-HEART Trial. Curr Cardiol Rep. 2016 Feb;18(2):18. doi: 10.1007/s11886-015-0695-4. PMID 26782999